CLINICAL TRIAL: NCT07159646
Title: Athletic Intervention After THoracic surgEry for luNg cAncer: a Pilot Study.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Collaborators: Università degli Studi di Pavia (Unknown)
Responsible Party: Principal Investigator, Giulia Maria Stella, Giulia Maria Stella, Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ATHENA study
Record Dates: First submitted 2025-08-26; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Non-small Cell Lung Cancer (NSCLC)
Keywords: NSCLC; athletic protocol; pulmonary function; HRQoL
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: Low risk, inactive non-invasive devices
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- athletic programs for NSCLC resected patients with good performance status (Experimental): evaluation procedures aimed at investigating exercise capacity, respiratory capacity and muscle power
  Interventions: Other: exercise interventions

INTERVENTIONS:
Other: exercise interventions — athletic/physical protocol

SUMMARY:
This is a pilot trial, monocentric interventional study that aims to investigate the results obtained by administering a specific athletic/physical protocol to a cohort of patients who undergo lung surgery after Non-small cell lung cancer (NSCLC) diagnosis.

Several studies explored the effects of combined aerobic and resistance training and demonstrated that exercise training improved fitness level (distance walked on the six-minute walk test) and which may also positively influence long-term HRQoL, fatigue, and exercise capacity. Due to the limited number of studies, the effect of exercise training on improvement of pulmonary function (FEV1 and DLCO) and quality of life and other outcomes is still unclear.

Several studies explored the effects of combined aerobic and resistance training, however few and controversial data are till now available regarding athletic programs for NSCLC resected patients with good performance status.

Ten consecutive patients who underwent resective surgery for NSCLC (5 males and 5 females) will be recruited in to the study.

Before and after the training program, patients will undergo evaluation procedures aimed at investigating exercise capacity, respiratory capacity and muscle power. Both the evaluations and exercise sessions will take place at the CRIAMS Sports Medicine Centre (University of Pavia).

Each patient will be addressed to a 6-month athletic program under the supervision of a motor scientist to evaluate if this active intervention could positively impact on the recovery and improvement of pulmonary function as well as on quality of life after surgery for cancer.

The primary endpoint will be the change of pulmonary function VO2 max) measured at baseline and at the 6 th month of the study. It is defined as the amount of oxygen consumed while sitting at rest and is equal to 3.5 ml O2 per kg body weight x min.

Study findings will be compared to storage data on NSCLC patients (with comparable features) who underwent surgery in absence of subsequent active training programs.

DETAILED DESCRIPTION:
The aim of this pilot study is to assess in a preliminary cohort the effect of an active athletic training program in improving respiratory function parameters as well as quality of life after resective surgery for lung cancer. Ten patients (5 males and 5 females) who underwent lung resection for cancer will be identified and selected based on their high PS, the absence of comorbidity and need of adjuvant therapy based on post operative TNM disease stage IA and after multidisciplinary evaluation by GINT. The study will last 6 months for each of the 10 subjects enrolled during 12 months. The subsequent follow up for each patient will last 6 months. Each patient will be addressed to a 6-month athletic program under the supervision of a motor scientist to evaluate if this active intervention could positively impact on the recovery and improvement of pulmonary function as well as on quality of life after surgery for cancer. Moreover, although a pilot study, we will also evaluate stratify patients based on their gender and age to evaluate potential impact of demographic features.

Study participants will be recruited at Fondazione IRCCS Policlinico San Matteo, SC Pneumologia among those patients affected by lung cancer and addressed to surgery with a curative setting. After surgery each case will be rediscussed multidisciplinary and patients with higher performance status, defined by ECOG score 0 and CCI score from 1 to 4, will be selected for the study.

Specifically the ECOG Performance Status Scale describes a patient's level of functioning in terms of their ability to care for themselves, daily activity, and physical ability. An ECOG score of 0 identifies a fully active person, able to perform all pre-disease services without limitations. The Charlson Comorbidity Index (CCI) is used to classify comorbid conditions which may influence mortality risk. The severity of comorbidity from mild (CCI scores of 1-2) to moderate (CCI scores of 3-4) is used for the selection of patients in the study. Higher scores indicate a more severe condition and consequently, a worse prognosis.

Data obtained will be compared to storage data and published ones on patients with the same features of those enrolled in the study, who are addressed on to follow up after surgery.

Patients will be followed by motor scientists during their active training. Exercises could be slightly modified and each modification will be reported to CRF. In case of need of relevant modification of the training exercises the patient will leave the study.

The patient will enter the study 30 days after surgery. The first screening visit will encompass spirometry, DLCO analysis and VO2 max calculation. Patients will also undergo electrocardiogram (ECG) as per clinical practice, standard routine blood exam and clinical visit. Then the patient will enter the trial and subsequent controls, similar to the first one will be done at 3rd and 6th month, at the end of the program. At the same intervals a total body CT scan will be performed, as per clinical practice. After the end of the active interventional study, patients will continue the standard follow up procedures according to national and international guidelines.

The primary endpoint will be the change of pulmonary function VO2 max) measured at baseline and at the 6 th month of the study. It is defined as the amount of oxygen consumed while sitting at rest and is equal to 3.5 ml O2 per kg body weight x min.

Secondary endpoint will be:

* the change of pulmonary function (FEV1 and DLCO and VO2 max) measured at baseline, at the 3 rd and at the 6 th month of the study. The latter is defined as the amount of oxygen consumed while sitting at rest and is equal to 3.5 ml O2 per kg body weight x min.
* The quality of life will be assessed by the EORTC QLQ-C30 (vers. 3) Questionnaire a 30-item instrument designed to measure quality of life in all cancer patients [21].
* Improvement in caloric consumption measured by metabolic equivalents (MET).

Although being a pilot study, demographic exploratory outcomes would be assessed. Results will be analysed to evaluate if observed differences in outcomes could be related to gender and/or age of the subjects since it is conceivable that the two variables could affect athletic performances and primary and secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female ≥18 years old
2. Patient underwent a curative surgical treatment of NSCLC (stage IA according to AIOM guidelines, website https://www.iss.it/documents/20126/8403839/LG149_Polmone_agg2024.pdf/9e22916b-799c-3966-7dc9-01762112ce94?version=1.0&t=1732534604319)
3. First whole body CT scan after surgery (executed according to routine procedures two months after surgery) negative for cancer recurrence
4. Patients highest scores of performance status, defined after multidisciplinary evaluation by Interdisciplinary Group for Tho-racic Neoplasms (GINT) using ECOG Performance Status Scale and Charlson Comorbidity Index (CCI). Subject with ECOG score 0 and CCI score from 1 to 4 is eligible.
5. Informed Consent as documented by signa-ture

Exclusion Criteria:

1. Requirement of adjuvant treatment
2. Women who are pregnant or breast feeding
3. Intention to become pregnant during the course of the study,
4. Lack of safe contraception, defined as: Female participants of childbearing potential, not using and not willing to continue using a medically reliable method of contraception for the en-tire study duration, such as oral, injectable, or implantable contraceptives, or intrauterine contraceptive devices, or who are not using any other method considered sufficiently reliable by the investigator in individual cases. (Female participants who are surgically sterilised/hysterectomised or post- meno-pausal for longer than 2 years are not considered as being of child bearing potential)
5. Other clinically significant concomitant disease states (e.g., respiratory failure, COPD, interstitial lung disease, hepatic dysfunction, cardiovascular disease)
6. Known or suspected non-compliance, drug or alcohol abuse,
7. Inability to follow the procedures of the study
8. Participation in another study with investigational asset within the 30 days preceding and during the present study
9. Enrolment of the investigator, his/her family members, em-ployees and other dependent persons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Primary endpoints will be improvement of pulmonary function (VO2max) | From enrollment to the 6 th month of the study
  The primary endpoint will be the change of pulmonary function (VO2 max) measured at baseline and at the 6 th month of the study. It is defined as the amount of oxygen consumed while sitting at rest and is equal to 3.5 ml O2 per kg body weight x min

CONTACTS AND LOCATIONS:
Overall Officials: Angelo Guido Corsico, MD,, Study Director — Fondazione IRCCS Policlinico San Matteo
Locations (1):
- Fondazione IRCCS Policlinico San Matteo di Pavia, Pavia, Pavia, Italy

REFERENCES:
- [Background] Omiya K, Itoh H, Osada N, Kato M, Koike A, Sagara K, Aoki K, Fu LT, Watanabe H, Kato K, Tanabe K, Murayama M. Impaired heart rate response during incremental exercise in patients with acute myocardial infarction and after coronary artery bypass grafting: evaluation of coefficients with Karvonen's formula. Jpn Circ J. 2000 Nov;64(11):851-5. doi: 10.1253/jcj.64.851. PMID 11110430
- [Background] Hinz A, Weis J, Faller H, Brahler E, Harter M, Keller M, Schulz H, Wegscheider K, Koch U, Geue K, Gotze H, Mehnert A. Quality of life in cancer patients-a comparison of inpatient, outpatient, and rehabilitation settings. Support Care Cancer. 2018 Oct;26(10):3533-3541. doi: 10.1007/s00520-018-4211-4. Epub 2018 Apr 26. PMID 29700655
- [Background] Saito H, Hatakeyama K, Konno H, Matsunaga T, Shimada Y, Minamiya Y. Impact of pulmonary rehabilitation on postoperative complications in patients with lung cancer and chronic obstructive pulmonary disease. Thorac Cancer. 2017 Sep;8(5):451-460. doi: 10.1111/1759-7714.12466. Epub 2017 Jul 11. PMID 28696575
- [Background] Voorn MJJ, Driessen EJM, Reinders RJEF, van Kampen-van den Boogaart VEM, Bongers BC, Janssen-Heijnen MLG. Effects of exercise prehabilitation and/or rehabilitation on health-related quality of life and fatigue in patients with non-small cell lung cancer undergoing surgery: A systematic review. Eur J Surg Oncol. 2023 Oct;49(10):106909. doi: 10.1016/j.ejso.2023.04.008. Epub 2023 May 2. PMID 37301638
- [Background] Yanagita Y, Arizono S, Tawara Y, Oomagari M, Machiguchi H, Tanahashi M, Katagiri N, Iida Y, Kozu R. Physical activity in patients with non-small cell lung cancer after lung resection. Clin Biomech (Bristol). 2024 May;115:106249. doi: 10.1016/j.clinbiomech.2024.106249. Epub 2024 Apr 13. PMID 38615547
- [Background] Huang CY, Hsieh MS, Hsieh PC, Wu YK, Yang MC, Huang SY, Tzeng IS, Lan CC. Pulmonary rehabilitation improves exercise capacity, health-related quality of life, and cardiopulmonary function in patients with non-small cell lung cancer. BMC Cancer. 2024 Feb 15;24(1):211. doi: 10.1186/s12885-024-11977-5. PMID 38360680
- [Background] Luo N, Dai F, Wang X, Hu B, Zhang L, Zhao K. Pulmonary Rehabilitation Exercises Effectively Improve Chronic Cough After Surgery for Non-small Cell Lung Cancer. Cancer Control. 2024 Jan-Dec;31:10732748241255824. doi: 10.1177/10732748241255824. PMID 38764164
- [Background] Ten Cate DWG, van den Berg R, Scholten-Bakker M, Molenaar CJL, von Meyenfeldt EM, Slooter GD, van den Broek FJC, Marres GMH. Multimodal prehabilitation in patients with non-small cell lung cancer: a feasibility study. J Thorac Dis. 2024 May 31;16(5):2776-2789. doi: 10.21037/jtd-23-1929. Epub 2024 May 10. PMID 38883662
- [Background] Balduyck B, Hendriks J, Lauwers P, Van Schil P. Quality of life evolution after surgery for primary or secondary spontaneous pneumothorax: a prospective study comparing different surgical techniques. Interact Cardiovasc Thorac Surg. 2008 Feb;7(1):45-9. doi: 10.1510/icvts.2007.159939. Epub 2007 Aug 17. PMID 17704125
- [Background] Zawadzka-Fabijan A, Fabijan A, Lochowski M, Pryt L, Polis B, Zakrzewski K, Kujawa JE, Kozak J. Functional and Disability Outcomes in NSCLC Patients Post-Lobectomy Undergoing Pulmonary Rehabilitation: A Biopsychosocial Approach. Cancers (Basel). 2024 Jun 20;16(12):2281. doi: 10.3390/cancers16122281. PMID 38927985
- [Background] Fevrier E, Yip R, Becker BJ, Taioli E, Yankelevitz DF, Flores R, Henschke CI, Schwartz RM; IELCART Investigators. Change in quality of life of stage IA lung cancer patients after sublobar resection and lobectomy. J Thorac Dis. 2020 Jul;12(7):3488-3499. doi: 10.21037/jtd-20-402. PMID 32802427
- [Background] Balduyck B, Hendriks J, Lauwers P, Van Schil P. Quality of life evolution after lung cancer surgery: a prospective study in 100 patients. Lung Cancer. 2007 Jun;56(3):423-31. doi: 10.1016/j.lungcan.2007.01.013. Epub 2007 Feb 16. PMID 17306905